CLINICAL TRIAL: NCT01980823
Title: Pre-Surgical "Window of Opportunity" Trial of the Combination of Metformin and Atorvastatin in Newly Diagnosed Operable Breast Cancer
Brief Title: Pre-Surgical Trial of the Combination of Metformin and Atorvastatin in Newly Diagnosed Operable Breast Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Katherine D. Crew, Associate Professor of Medicine and Epidemiology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAM2306
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer; Breast Tumors; Cancer of Breast
Keywords: Breast Cancer; Metformin; Atorvastatin; Ki-67
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin; Atorvastatin; Mastectomy, Segmental

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Metformin-Atorvastatin combination (Experimental): Patients will receive metformin and atorvastatin for approximately 2 weeks prior to breast surgery.
  Interventions: Drug: Metformin; Drug: Atorvastatin; Procedure: Breast surgery

INTERVENTIONS:
Drug: Metformin — Metformin is an oral diabetes medicine that helps control blood sugar levels.
  Dosage/Frequency: 1500 mg per day: divided 500 mg in the morning and 1000 mg in the evening
  Metformin is for people with type 2 diabetes. Metformin is sometimes used in combination with insulin or other medications, but it is not for treating type 1 diabetes.
  Other Names: Glucophage
Drug: Atorvastatin — Atorvastatin is in a group of drugs called "statins." Atorvastatin reduces levels of "bad" cholesterol (low-density lipoprotein, or LDL) and triglycerides in the blood while increasing levels of "good" cholesterol (high-density lipoprotein, or HDL).
  Dosage/Frequency: 80 mg once a day at bedtime
  Atorvastatin is used to treat high cholesterol, and to lower the risk of stroke, heart attack, or other heart complications in people with type 2 diabetes, coronary heart disease, or other risk factors.
  Other Names: Lipitor
Procedure: Breast surgery — (Non-experimental) Female subjects with histologically-confirmed operable invasive breast cancer or DCIS will undergo core needle biopsy with a plan of surgical excision.
  Other Names: No other name

SUMMARY:
The purpose of this study is to determine the effects of combining metformin and atorvastatin treatment in patients with newly diagnosed breast cancer during the interval between breast biopsy and surgery.

This study is designed to assess whether tumor proliferation, as measured by the natural log expression of Ki-67 staining of breast tumor cells, is reduced following approximately 2 weeks of treatment with the combination of metformin plus atorvastatin in patients with newly diagnosed breast cancer.

DETAILED DESCRIPTION:
Breast cancer cells require energy homeostasis shifts with enhanced anabolism to enable rapid growth and continued proliferation. The main energy regulatory system in eukaryotes and breast cancer cells is the AMP-activated kinase (AMPK) pathway. AMPK is triggered by changes in the AMP/Adenosine triphosphate (ATP) ratio thus impacting energy reserves and requirements. AMPK pathway closely interacts with the phosphoinositide 3-kinase (PI3K)/Akt signaling pathway, affecting the downstream function of the master regulator mammalian target of rapamycin (mTOR). Activation of AMPK has been shown in vitro to result in inhibition of proliferation of various cancer cell lines.

Utilizing a pre-surgical model, the investigator plans to conduct a pilot study of 40 women with newly diagnosed invasive breast cancer or ductal carcinoma in-situ (DCIS) who will receive oral metformin and atorvastatin daily in the interval between diagnostic breast biopsy and definitive breast surgery.

The goal is to determine if dual combination treatment with metformin plus atorvastatin significantly impacts tumor-based markers, such as proliferation, and blood-based biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects with histologically-confirmed operable invasive breast cancer or DCIS, who undergo core needle biopsy followed by surgical excision at least 2 weeks after enrollment
* ≥ 5 mm by imaging/pathology of core to ensure enough pre- and post-treatment tissue for analysis
* Age ≥ 21 years. Breast cancer is uncommon in patients less than this age.
* No prior chemotherapy, radiation therapy, or breast resection within 6 months of study entry
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Signed informed consent

Exclusion Criteria:

* Currently on medication for diabetes or hypercholesterolemia
* Treatment with other investigational drugs within 6 months of study entry
* Strong Cytochrome P450 3A4 (abbreviated CYP3A4) (e.g., clarithromycin, HIV protease inhibitors, and itraconazole), given potential interactions with atorvastatin
* Renal impairment with a creatinine > 1.4 mg/dl
* Hepatic impairment: Aspartate transaminase (AST)/(SGOT), Alanine Transaminase(ALT)/(SGPT) ≥ 2.5 x upper limit of normal range (ULN), OR Total bilirubin ≥ 1.5 x ULN (subjects with Gilbert's syndrome can have bilirubin of up to 1.5 x ULN), OR Alkaline phosphatase > 2.5 x ULN

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Change in tissue levels of the proliferation marker Ki-67 | Baseline, 2 weeks after start of treatment
  Tumor proliferation, as measured by the natural log expression of Ki-67 staining of breast tumor cells.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Crew, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center - Herbert Irving Cancer Center, New York, New York, United States

REFERENCES:
- See also: Herbert Irving Comprehensive Cancer Center (HICCC) Clinical Trials Page — https://cancer.columbia.edu/